CLINICAL TRIAL: NCT00849953
Title: FinESS Registry Study
Status: Completed | Type: Observational
Sponsor: Entellus Medical, Inc. (Industry)
Responsible Party: Entellus Medical, Entellus Medical
Other Study IDs: 1498-001
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FinESS Treatment: Subjects undergoing treatment with the FinESS Sinus Treatment System

SUMMARY:
A prospective, post-approval registry study assessing subject rhinosinusitis symptomatic status over time following treatment with FinESS Sinus Treatment using self-administered quality of life survey data.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 years or older undergoing balloon dilation with FinESS Sinus Treatment and have provided voluntary consent to participate in Registry

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who in the investigator's opinion, require trans-antral treatment of the maxillary sinus ostium and ethmoid infundibulum to remodel the bony sinus outflow tract using balloon displacement of adjacent bone and paranasal sinus structures using FinESS Sinus Treatment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Grebner, Study Director — Entellus Medical
Locations (14):
- United States (14):
  - South Denver ENT and Allergy, Denver, Colorado
  - Gulf Coast Facial Plastics and ENR, Panama City, Florida
  - Gensys Regional Medical Center, Grand Blanc, Michigan
  - Paparella Group, Maple Grove, Minnesota
  - St. Cloud Ear Nose and Throat, Saint Cloud, Minnesota
  - Lee's Summit Ear, Nose and Throat Center, Lee's Summit, Missouri
  - Midwest Ear, Nose and Throat, Sioux Falls, South Dakota
  - Dickson Ear, Nose and Throat PLC, Dickson, Tennessee
  - Austin Ear, Nose and Throat Clinic, Austin, Texas
  - Capital Otolaryngology, Austin, Texas
  - Texas Sinus Center, Boerne, Texas
  - Medical Center ENT Associates of Houston, Houston, Texas
  - Advanced Otolaryngology, PC, Richmond, Virginia
  - Advanced Ear, Nose and Throat Specialists, Milwaukee, Wisconsin